| Division | : Worldwide Development |
|------------------|-------------------------------|
| Information Type | : Reporting and Analysis Plan |

Title : Reporting and Analysis Plan for Study 204824: A Phase 2, Pilot, Multicenter, Single Arm Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of GSK1070806 plus Standard of Care for the Prevention of Delayed Graft Function in Adult Subjects After Renal Transplantation

Compound Number : GSK1070806

Effective Date : May-24-2017

## **Description:**

- The purpose of this Reporting and Analysis Plan (RAP) is to describe the planned efficacy, safety & tolerability, and pharmacokinetics analyses and output to be included in the Clinical Study Report for Protocol 204824.
- This document will be provided to the study team members to convey the content of interim and final Statistical Analysis Complete (SAC) deliverable.
- Purpose of RAP Amendment 1:
  - Change the number of patients for dose escalation interim analysis from 8 -10 to 6 to match the protocol amendment.
  - Remove outputs for the IA1 delivery which are no longer required for a dose escalation decision, defined as IA1 in this document.

#### **Author's Name and Functional Area:**

| PPD | May-24-2017 |
|-----------------------------------------------------------|--------------|
| Principal Statistician (Clinical Statistics) | May-24-2017 |
| PPD | May-24-2017 |
| Director (Clinical Pharmacology, Modeling and Simulation) | Wiay-24-2017 |
| PPD | May-24-2017 |
| Director (Quantitative Clinical Pharmacology), PAREXEL | Way-24-2017 |

## Approved by:

| PPD | May 24 2017 |
|--------------------------------------------------|-------------|
| Senior Statistics Director (Clinical Statistics) | May-24-2017 |


## The GlaxoSmithKline group of companies

204824

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| 1. | REPORTING & ANALYSIS PLAN SYNPOSIS | 5 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 6 |
| 4. | 2.1. Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. Study Objective(s) and Endpoint(s) | 6 |
| | 2.3. Study Design | |
| | 2.4. Statistical Hypotheses | |
| | 2.5. Definition of Renal Graft Function | |
| | | , |
| 3. | PLANNED ANALYSES | 9 |
| | 3.1. Interim Analyses | |
| | 3.2. Final Analyses | 10 |
| 4. | ANALYSIS POPULATIONS | 12 |
| | 4.1. Protocol Deviations | 12 |
| 5. | GENERAL CONSIDERATIONS FOR DATA ANALYSES AND DATA | 12 |
| | HANDLING CONVENTIONS | 13 |
| 6. | STUDY POPULATION ANALYSES | 13 |
| | 6.1. Planned Analyses Overview | 13 |
| 7 | DDIMADY OTATIOTICAL ANALYCEO | 1.4 |
| 7. | PRIMARY STATISTICAL ANALYSES | |
| | 7.1. Final Analyses | 13 |
| 8. | SECONDARY STATISTICAL ANALYSES | 14 |
| | 8.1. Efficacy Analyses | |
| | 8.1.1. Overview of Planned Efficacy Analyses | |
| | 8.1.2 AUC and 1/2 Life Time. | |
| | 8.2. Safety Analyses | |
| | 8.2.1. Overview of Planned Analyses | |
| | 8.3. Pharmacokinetic Analyses. | |
| | 8.3.1. Overview of Planned Pharmacokinetic Analyses | |
| | 8.3.2. Drug Concentration Measures | |
| | 8.3.3. Pharmacokinetic Parameters | |
| | 8.3.3.1. Deriving Pharmacokinetic Parameters | |
| 0 | OTHER CTATICTICAL ANALYCES | 200 |
| 9. | OTHER STATISTICAL ANALYSES 9.1. Overview of Planned Pharmacokinetic / Pharmacodynamic Analyses | |
| | 9.1. Overview of Flatined Flatinacokinetic / Flatinacodynamic Analyses | 19 |
| 10. | REFERENCES | 21 |
| 11. | APPENDICES | |
| | 11.1. Appendix 1: Protocol Deviation Definitions for Per Protocol Population | |
| | 11.2. Appendix 2: Time and Events | |
| | 11.3. Appendix 3: Treatment States and Phases | |
| | 11.3.1. Treatment Phases | |
| | 11.3.2 Treatment States | 287 |


## GSK1070806

| | 11.3.3. | Treatment States for AE Data | <mark>28</mark> 7 |
|---|---|---|---|
| 11.4. | Appendix | 4: Data Display Standards & Handling Conventions | |
| | 11.4.1. | Baseline Definition & Derivations | |
| | | 11.4.1.1. Baseline Definitions | 29 |
| | | 11.4.1.2. Derivations and Handling of Missing Baseline Data | 29 |
| | 11.4.2. | Reporting Process & Standards | 29 |
| 11.5. | Appendix | 5: Derived and Transformed Data | 321 |
| | 11.5.1. | General | 321 |
| | 11.5.2. | Study Population | 321 |
| | 11.5.3. | Safety | |
| 11.6. | Appendix | 6: Premature Withdrawals & Handling of Missing Data | 34 |
| | 11.6.1. | Premature Withdrawals | |
| | 11.6.2. | Handling of Missing Data | 344 |
| | | 11.6.2.1. Handling of Missing Dates | 344 |
| | | 11.6.2.2. Handling of Partial Dates | 355 |
| 11.7. | Appendix | 7: Values of Potential Clinical Importance | 376 |
| | 11.7.1. | Laboratory Values | 376 |
| | 11.7.2. | ECG | 387 |
| | 11.7.3. | Vital Signs | 387 |
| 11.8. | Appendix | 8 – Abbreviations & Trade Marks | 38 |
| | 11.8.1. | Abbreviations | 38 |
| | 11.8.2. | Trademarks | 39 |
| 11.9. | Appendix | 9: List of Data Displays | 40 |
| | 11.9.1. | Data Display Numbering | 40 |
| | 11.9.2 | Deliverable | 40 |
| | 11.9.3. | Study Population Tables | 41 |
| | 11.9.4. | Efficacy Tables | 43 |
| | 11.9.5. | Efficacy Figures | 49 |
| | 11.9.6. | Safety Tables | 50 |
| | 11.9.7. | Pharmacokinetic Tables | 54 |
| | 11.9.8. | Pharmacokinetic Figures | 55 |
| | 11.9.9. | Pharmacokinetic / Pharmacodynamic Figures | |
| | 11.9.10. | ICH Listings | 56 |
| | 11.9.11. | Non-ICH Listings | |
| 11.10. | Appendix | 10: Example Mock Shells for Data Displays | 64 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Purpose This RAP details all planned analyses and outputs required for the final Clin Study Report (CSR) of study 204824. Protocol This RAP is based on the protocol (Dated: 03-FEB-2016 for study 204824 [GlaxoSmithKline Document Number: 2015N240632_01]. Primary Objective Evaluate the efficacy of single intravenous dose administrations of GSK 1070806 in prevention of delayed graft function (DGF) after transplantation. Primary Endpoint Primary Analysis Population Public This RAP details all planned analyses and outputs required for the final Clin Study 204824 [GlaxoSmithKline Document Number: 2015N240632_01]. Primary Endpoint Proportion of single intravenous dose administrations of GSK 1070806 in prevention of delayed graft function (DGF) after transplantation. Primary Analysis Population | |
|---|---|
| Primary Objective | cal |
| <ul> <li>Primary Objective</li></ul> | |
| Objective GSK1070806 in prevention of delayed graft function (DGF) after transplantation. Primary Endpoint Proportion of subjects requiring dialysis during the first 7 days post transplat (excluding requirement for dialysis due to hyperkalemia within first 24 post-operative hours). Study Design Pilot, multicenter, single arm Bayesian sequential design study to evaluate the efficacy, safety, tolerability and pharmacokinetics (PK) of GSK1070806 in patients undergoing renal transplantation. Sample size (maximum of 30) had been selected to yield the probability of a "go" decision of 0.139 when the GSK1070806 DGF rate is 50% and 0.69 at what has been considered to be a clinically impactful GSK1070806 DGF rate 35%. Planned Analyses Interim analyses are detailed within Section 3.1 where applicable. All decisions regarding final analysis, as defined in this RAP document, will made prior to Database Freeze of the study data. Primary Analysis Population The 'Analysis Population' will be used to evaluate DGF related endpoints The 'All Subjects Population' will be used to evaluate study population; safe PD/Biomarkers and other efficacy endpoints. | |
| <ul> <li>Endpoint (excluding requirement for dialysis due to hyperkalemia within first 24 post-operative hours).</li> <li>Study Design Pilot, multicenter, single arm Bayesian sequential design study to evaluate the efficacy, safety, tolerability and pharmacokinetics (PK) of GSK1070806 in patients undergoing renal transplantation.</li> <li>Sample size (maximum of 30) had been selected to yield the probability of a "go" decision of 0.139 when the GSK1070806 DGF rate is 50% and 0.69 at what has been considered to be a clinically impactful GSK1070806 DGF rate 35%.</li> <li>Planned Analyses Interim analyses are detailed within Section 3.1 where applicable.</li> <li>All decisions regarding final analysis, as defined in this RAP document, will made prior to Database Freeze of the study data.</li> <li>Primary Analysis Population Will be used to evaluate DGF related endpoints</li> <li>The 'Analysis Population' will be used to evaluate study population; safe PD/Biomarkers and other efficacy endpoints.</li> </ul> | |
| <ul> <li>efficacy, safety, tolerability and pharmacokinetics (PK) of GSK1070806 in patients undergoing renal transplantation.</li> <li>Sample size (maximum of 30) had been selected to yield the probability of a "go" decision of 0.139 when the GSK1070806 DGF rate is 50% and 0.69 at what has been considered to be a clinically impactful GSK1070806 DGF rate 35%.</li> <li>Planned Analyses</li> <li>Interim analyses are detailed within Section 3.1 where applicable.</li> <li>All decisions regarding final analysis, as defined in this RAP document, will made prior to Database Freeze of the study data.</li> <li>Primary Analysis Population' will be used to evaluate DGF related endpoints</li> <li>The 'Analysis Population' will be used to evaluate study population; safe PD/Biomarkers and other efficacy endpoints.</li> </ul> | it |
| <ul> <li>"go" decision of 0.139 when the GSK1070806 DGF rate is 50% and 0.69 at what has been considered to be a clinically impactful GSK1070806 DGF rate 35%.</li> <li>Planned Analyses</li> <li>Interim analyses are detailed within Section 3.1 where applicable.</li> <li>All decisions regarding final analysis, as defined in this RAP document, will made prior to Database Freeze of the study data.</li> <li>Primary Analysis Population' will be used to evaluate DGF related endpoints</li> <li>The 'Analysis Population' will be used to evaluate study population; safe PD/Biomarkers and other efficacy endpoints.</li> </ul> | e |
| Analyses Analyses Analyses All decisions regarding final analysis, as defined in this RAP document, will made prior to Database Freeze of the study data. Primary Analysis Population The 'Analysis Population' will be used to evaluate DGF related endpoints The 'All Subjects Population' will be used to evaluate study population; safe PD/Biomarkers and other efficacy endpoints. | e of |
| Primary Analysis Population A | |
| Analysis Population The 'All Subjects Population' will be used to evaluate study population; safe PD/Biomarkers and other efficacy endpoints. | be |
| Population PD/Biomarkers and other efficacy endpoints. | |
| | ty; |
| • The 'PK' population will be used to evaluate pharmacokinetics. | |
| • The 'Per-Protocol' population will be used to evaluate the DGF rate in addit to the 'Analysis Population'. | on |
| Hypothesis • The study is to determine the effect of GSK1070806 on DGF. Stopping rule have been defined to test whether the DGF rate is less than or equal to the number hypothesis rate of 50%. | |
| Primary • A summary of the observed DGF rate during the study will be provided. | |
| • The posterior probability that the proportion of subjects experiencing DGF i less than 50% will be calculated. | ' |
| Secondary Analyses Summaries of baseline and post-dose values or proportions of subjects at various time points will be provided. | |
| Graft survival will be summarized by Kaplan-Meier plots. | |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Not applicable.

# 2.2. Study Objective(s) and Endpoint(s)

| Obj | jectives | Endpoints |
|---|---|---|
| | mary | Primary |
| • | To assess the frequency of delayed graft function (DGF) in donation after circulatory death (DCD) renal transplant recipients treated with GSK1070806. | • Proportion of subjects requiring dialysis during the first 7 days post transplant, (excluding requirement for dialysis due to hyperkalemia within first 24 post-operative hours). |
| Sec | ondary | Secondary |
| • | To assess graft function in DCD renal transplant recipients treated with GSK1070806. | <ul> <li>Serum creatinine at baseline and over time post transplant.</li> <li>Urine output at baseline and over time post transplant.</li> <li>Proportion of subjects in the first 7 days with:</li> </ul> |
| | | <ul> <li>Primary Non Function</li> <li>Functional DGF</li> <li>Intermediate Graft Function</li> <li>Immediate Graft Function</li> </ul> |
| • | To assess the effect of GSK1070806 on acute rejection risk, and rejection/PD biomarkers. | <ul> <li>Proportion of subjects with episodes of biopsy-proven acute rejection.</li> <li>Rejection biomarkers/ PD markers (including serum IP-10 and Mig) at baseline and over time post transplant.</li> </ul> |
| • | To assess the effect of GSK1070806 on dialysis dependency and graft survival. | <ul> <li>Number of dialysis events per patient in the first 30 days post transplant.</li> <li>Proportion of subjects who are dialysis-independent at visits up to 12 months post transplant.</li> </ul> |
| • | To assess the safety and tolerability of GSK1070806 in renal transplant recipients. | <ul> <li>AEs and SAEs</li> <li>Clinical laboratory values</li> <li>Vital signs</li> <li>Frequency, type and severity of infections</li> </ul> |
| • | To assess the pharmacokinetics of GSK1070806 in renal transplant recipients. | Serum concentrations of GSK1070806 over<br>time, and derived pharmacokinetic<br>parameters if feasible (AUC, Cmax). |

| Objectives | Endpoints |
|---|---|
| To assess the effect of<br>GSK1070806 administration on<br>serum IL-18 levels. | • Free, total, and GSK1070806 bound IL-18 at baseline and over time post transplant. |
| To determine immunogenicity of<br>GSK1070806 in renal transplant<br>recipients. | <ul> <li>Frequency of anti-drug antibodies (ADAs) before and after GSK1070806 administration.</li> <li>ADA titers.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Exploratory | Exploratory |
| To assess the impact of<br>GSK1070806 on urine biomarkers<br>of renal injury. | • Serial measurements of urinary biomarkers, including KIM-1, NGAL and IL-18, at baseline and over time post transplant. |
| To assess IL-18 target engagement in the kidney. | GSK1070806 and IL-18 levels within renal graft biopsies, as assessed by immunohistochemistry. |
| • To assess the relation between IL-<br>18 levels in renal preservation<br>fluid and graft function. | Level of IL-18 in renal preservation fluid. |
| To assess the impact of<br>GSK1070806 administration on<br>IL-18 binding protein levels. | Serum IL-18 binding protein at baseline and over time post transplant. |
| To assess the humoral and cellular response to the transplanted organ | Serum cytokine levels at baseline and over time post transplant. |
| in the presence of GSK1070806. | Histological analysis of biopsies with respect to cellular infiltrate. |
| To assess health outcomes in | Length of hospital stay |
| renal transplant recipients following GSK1070806 administration. | Re-hospitalization |

## 2.3. Study Design



## 2.4. Statistical Hypotheses

The study is to determine the effect of GSK1070806 on DGF. Stopping rules have been defined to test whether the DGF rate is less than or equal to the null hypothesis rate of 50%.

#### 2.5. Definition of Renal Graft Function

## **Primary Non Function:**

• Permanent lack of function of the allograft defined as an inability to discontinue dialysis from the time of transplantation. Note: The study site will decide whether patients have primary non function DGF or not and record it in data set.

## 3 day Functional Delayed Graft Function:

• <10% fall in SCr versus baseline per day averaged over first 3 days with OR without dialysis

## 7 day Functional Delayed Graft Function:

• <30% reduction in baseline SCr in first 7 days with OR without dialysis

#### 3 day Intermediate Graft Function:

• 10-20% fall in SCr versus baseline per day averaged over first 3 days without dialysis

#### 7 day Intermediate Graft Function:

• 30-70% reduction in baseline Cr in first 7 days without dialysis

#### 3 day Immediate Graft Function:

• >20% fall in SCr versus baseline per day averaged over first 3 days without dialysis

## 7 day Immediate Graft Function:

• >70% reduction in baseline Cr during the first 7 days without dialysis

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

## 3.1.1 Bayesian Sequential Analysis

The DGF data will be reviewed sequentially. The sequential decision rule is shown graphically in Figure 1. The number in the first column indicates the number of subjects who have completed study treatment. From the point in time when approximately 6 subjects have reached day 7 post transplantation the sponsor study team will begin to evaluate the DGF rates. This will start with the first 6 subjects and then with addition of data from each subsequent subject that completes 7 days of the trial. A sequential Go/No Go/Continue rule is based on the predictive probability of success. A high predictive probability (PP) of success means that GSK1070806 is likely to be efficacious by the end of the study given the observed data, whereas a low PP suggests that the treatment may not have sufficient activity. If the PP value is less than 2% (red region) the trial may be stopped and the alternative hypothesis will be rejected. If the PP is greater 92% (green), the conclusion may be made that GSK1070806 has better efficacy than the standard of care. If the PP is between 2 - 92% (white region), the trial will continue to the next interim analysis (to be conducted after the next subject has completed treatment) or until reaching 30 completed subjects.

## 3.1.2 Planned Interim Analysis

The following interim analyses are planned (protocol defined):

| Interim | Details |
|---|---|
| Analysis | |
| During<br>Study | <ul> <li>The DGF data will be reviewed sequentially.</li> <li>An interim analysis will be performed after recruitment of approximately 8 to 10 patients to review for a consideration of dose adjustment based on an integrated review of safety/tolerability, efficacy, and exposure.</li> <li>The preliminary PK data which involves but not limited to GSK1070806 concentrations, total, free, drug bound IL-18 levels as data permit and applicable.</li> <li>Once the last patient completes 7-Days post-transplant, an interim analysis will be performed of all available data for the primary endpoint in addition to supportive efficacy and safety data. The results of this interim analysis will be reviewed by the GSK study team and other relevant GSK staff for internal decision making.</li> </ul> |

# 3.2. Final Analyses

A summary of the observed DGF rate during the study will be provided. The posterior probability that the proportion of subjects experiencing DGF is less than 50% will be calculated.

Figure 1 Sequential Decision Rules

# # DGF Events

| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 0.515 | | | | | | | | | | | | |
| | 1 | 0.618 | 0.35 | | | | | | | | | | | |
| | 2 | 0.71 | 0.452 | 0.215 | | | | | | | | | | |
| | 3 | 0.788 | 0.553 | 0.3 | 0.119 | | | | | | | | | |
| | 4 | 0.852 | 0.649 | 0.394 | 0.179 | 0.058 | | | | | | | | |
| | 5 | 0.9 | 0.735 | 0.492 | 0.253 | 0.095 | 0.025 | | | | | | | |
| | 6 | 0.936 | 0.808 | 0.589 | 0.339 | 0.146 | 0.045 | 0.009 | | | | | | |
| | 7 | 0.961 | 0.867 | 0.68 | 0.433 | 0.21 | 0.074 | 0.018 | 0.003 | | | | | |
| | 8 | 0.977 | 0.912 | 0.761 | 0.53 | 0.288 | 0.116 | 0.033 | 0.006 | 8E-04 | | | | |
| | 9 | 0.988 | 0.945 | 0.83 | 0.624 | 0.376 | 0.17 | 0.055 | 0.012 | 0.002 | 2E-04 | | | |
| $\overline{\mathbf{o}}$ | 10 | 0.994 | 0.967 | 0.884 | 0.712 | 0.47 | 0.239 | 0.088 | 0.023 | 0.004 | 4E-04 | 2E-05 | | |
| Evaluated | 11 | 0.997 | 0.982 | 0.926 | 0.79 | 0.567 | 0.32 | 0.133 | 0.039 | 0.008 | 9E-04 | 6E-05 | 1E-06 | |
| 3 | 12 | 0.999 | 0.991 | 0.955 | 0.854 | 0.661 | 0.411 | 0.192 | 0.064 | 0.014 | 0.002 | 1E-04 | 4E-06 | 0 |
| Š | 13 | 0.999 | 0.996 | 0.975 | 0.905 | 0.747 | 0.508 | 0.265 | 0.1 | 0.025 | 0.004 | 3E-04 | 1E-05 | 0 |
| | 14 | 1 | 0.998 | 0.987 | 0.942 | 0.821 | 0.606 | 0.351 | 0.148 | 0.043 | 0.008 | 8E-04 | 3E-05 | 0 |
| 뜓 | 15 | 1 | 0.999 | 0.994 | 0.967 | 0.881 | 0.7 | 0.447 | 0.212 | 0.069 | 0.014 | 0.002 | 8E-05 | 0 |
| Patients | 16 | 1 | 1 | 0.998 | 0.983 | 0.927 | 0.785 | 0.548 | 0.29 | 0.107 | 0.025 | 0.003 | 2E-04 | 0 |
| ā | 17 | 1 | 1 | 0.999 | 0.992 | 0.959 | 0.856 | 0.65 | 0.382 | 0.159 | 0.043 | 0.006 | 4E-04 | 0 |
| # - | 18 | 1 | 1 | 1 | 0.997 | 0.98 | 0.912 | 0.745 | 0.485 | 0.228 | 0.07 | 0.012 | 9E-04 | 0 |
| | 19 | 1 | 1 | 1 | 0.999 | 0.991 | 0.951 | 0.828 | 0.593 | 0.314 | 0.109 | 0.022 | 0.002 | 0 |
| | 20 | 1 | 1 | 1 | 1 | 0.997 | 0.977 | 0.895 | 0.7 | 0.415 | 0.165 | 0.038 | 0.004 | 0 |
| | 21 | 1 | 1 | 1 | 1 | 0.999 | 0.991 | 0.944 | 0.798 | 0.529 | 0.24 | 0.063 | 0.007 | 0 |
| | 22 | 1 | 1 | 1 | 1 | 1 | 0.997 | 0.975 | 0.879 | 0.649 | 0.336 | 0.102 | 0.013 | 0 |
| | 23 | 1 | 1 | 1 | 1 | 1 | 1 | 0.992 | 0.939 | 0.764 | 0.454 | 0.161 | 0.024 | 0 |
| | 24 | 1 | 1 | 1 | 1 | 1 | 1 | 0.998 | 0.977 | 0.864 | 0.587 | 0.245 | 0.044 | 0 |
| | 25 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0.995 | 0.939 | 0.725 | 0.359 | 0.077 | 0 |
| | 26 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0.984 | 0.854 | 0.505 | 0.134 | 0 |
| | 27 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0.951 | 0.679 | 0.226 | 0 |
| | 28 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0.861 | 0.377 | 0 |
| | 29 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0.619 | 0 |
| | 30 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 |

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | <b>Analyses Evaluated</b> |
|---|---|---|
| All Subjects | • Comprise of subjects who receive the dose of | • Safety/tolerability |
| | study medication. | |
| Analysis | For DGF related endpoints the 'Analysis | <ul> <li>Efficacy</li> </ul> |
| _ | Population' (AP) is defined as subjects in the | <ul> <li>PD/Biomarker</li> </ul> |
| | 'All Subjects' population who have been | |
| | declared to have DGF or have reached 7 days. | |
| | For other endpoints, the AP is defined as | |
| | subjects having baseline and at least one post- | |
| | baseline assessment. | |
| Per | Comprised of Analysis Population subjects who | <ul> <li>Primary efficacy</li> </ul> |
| Protocol | are compliant with protocol-specific criteria. | endpoint |
| | Subjects with specified protocol deviations will | |
| | be excluded per Appendix 1. | |
| PK | • Subjects in the 'All Subjects' population for | • PK |
| | whom a serum pharmacokinetic sample is | |
| | obtained and analyzed for GSK1070806. | |

#### **NOTE:**

• Please refer to Appendix 10: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Definitions for Per Protocol Population).
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - O Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. GENERAL CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

• There are no planned adjustments made for multiple centres in this study.

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 11.1 | Appendix 1: Protocol Deviation Definitions for Per Protocol Population |
| 11.2 | Appendix 2: Time and Events |
| 11.3 | Appendix 3: Treatment States and Phases |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |
| Error!<br>Referenc<br>e source<br>not<br>found. | : Laboratory A&R (QUEST: LAB) Dataset Details |
| Error!<br>Referenc<br>e source<br>not<br>found. | Appendix 1: Abbreviations |
| 11.10 | Appendix 10: List of Data Displays |
| 11.11 | Appendix 11: Mock Data Displays |

## 6. STUDY POPULATION ANALYSES

## **6.1.** Planned Analyses Overview

The study population analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses with full details of data displays being presented in Appendix 11.10: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| | Figure | Table | Listing |
|---|---|---|---|
| <b>Subject Disposition</b> | | | |
| Subject Disposition | | Y | |
| Reasons for Screening Failures | | Y | Y |
| Reasons for Withdrawals | | Y | Y |
| Important Protocol Deviations | | | Y |
| Deviations Leading to Exclusions from PP<br>Population | | | Y |
| Inclusion and Exclusion Criteria Deviations | | | Y |
| Demography (recipient) | | | |
| Demographics Characteristics | | Y | Y |
| Race & Racial Combinations | | Y | Y |
| Study Populations | | Y | Y [1] |
| Medical Condition & Concomitant Medication | ns | | |
| Medical Conditions (Current/Past) | | Y | Y |
| Concomitant Medication | | Y | Y |
| Virology (recipient) | | | Y |
| Donor Kidney Data | | | |
| Virology (donor) | | | Y |
| Demography (donor) | | Y | Y |
| Characteristics (donor) | | | Y |

#### **NOTES:**

## 7. PRIMARY STATISTICAL ANALYSES

A summary of the observed DGF rate during the study will be provided. The observed DGF rate will be calculated based on "Analysis" population as the primary analysis and based on "Per Protocol" population as sensitivity analysis.

## 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Efficacy Analyses

## 8.1.1. Overview of Planned Efficacy Analyses

The secondary efficacy analyses will be based on the "Analysis" population, unless otherwise specified.

<sup>1.</sup> Listing of subjects excluded from any population will be generated only.

Table 3 provides an overview of the planned efficacy analyses with further details of data displays being presented in Appendix 11.10: List of Data Displays.

Table 3 Overview of Planned Efficacy Analyses

| Endpoints | | Abso | olute | | C | hange fro | m Baseli | ne |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Indi | vidual | Sum | Summary | | Individual |
| | Т | F | F | L | Т | F | F | L |
| Graft function | | | | 1 | | | | l |
| Serum creatinine | Y | Y | Y | Y | Y | Y | Y | Y |
| Creatinine - AUC | Y | | | Y | | | | |
| Creatinine – ½ life | Y | | | Y | | | | |
| Urine output | | | Y | Y | | | | Y |
| Primary Non<br>Functions | Y | | | Y | | | | |
| Functional DGF | Y | | | Y | | | | |
| Intermediate graft function | Y | | | Y | | | | |
| Immediate graft function | Y | | | Y | | | | |
| Acute rejection risk a | ınd rejec | tion/PD b | iomarke | r | | | | |
| Episode of biopsy-<br>proven acute<br>rejection | Y | | | Y | | | | |
| Serum IP-10 | Y | Y | Y | | Y | Y | Y | |
| Serum Mig | Y | Y | Y | | Y | Y | Y | |
| Serum IL-18 levels | | | | | | | , | , |
| Free IL-18 | Y | Y | Y | | Y | Y | Y | |
| Bound IL-18 | Y | Y | Y | | Y | Y | Y | |
| Total IL-18 | Y | Y | Y | | Y | Y | Y | |
| Urine biomarkers | | T | T | T | | ı | T | r |
| IL-18 | Y | Y | | Y | | | | |
| NGAL | Y | Y | | Y | | | | |
| KIM1 | Y | Y | | Y | | | | |
| Dialysis dependency | and graft | survival | T | 1 | | T | 1 | 1 |
| Number of dialysis<br>events per patient in<br>the first 30 days post<br>transplant | Y | | | Y | | | | |
| Proportion of<br>subjects who are<br>dialysis-independent<br>at visits up to 12<br>months post<br>transplant | Y | | | | | | | |

| Exploratory | | | | | | |
|---|---|---|---|---|---|---|
| % free GSK1070806<br>within renal graft<br>biopsies | Y | | Y | | | |
| % bound<br>GSK1070806 within<br>renal graft biopsies | Y | | Y | | | |
| Level of IL-18 in<br>renal preservation<br>fluid | Y | | Y | | | |
| Serum IL-18 binding protein | | Y | | | | |
| Serum cytokine levels | Y | Y | | Y | Y | |
| Histological analysis of biopsies with respect to cellular infiltrate | | | | | | Y |
| Length of hospital stay | Y | | Y | | | |
| Re-hospitalization | | | Y | | | |

#### **NOTES:**

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 8.1.2. AUC and ½ Life Time

For serum creatinine, the 7-Day Area under the Curve (AUC), 30-Day AUC and 30 Day ½ life time will be calculated. The formula to calculate the AUC is:

 $AUC = \sum_{i=1}^{M} 1/2(Y_i + Y_{i-1})(d_i - d_{i-1})$  where  $Y_i$  is the serum creatinine value at Day  $d_i$  and M is the total number of measures the patient has. The 7 Day AUC will be calculated based on patients who have serum creatinine value at Day 7. The patients who will be discharged before Day 7 will be excluded from calculation. All patients are expected to have serum creatinine 30 Day post transplant. If the value is missing, the patient will be excluded from calculation.

The algorithm to determine the ½ life time is:

1. Determine the  $\frac{1}{2}$  value by  $Y_{1/2} = \frac{1}{2} * Y_0$  where  $Y_0$  is the baseline value for non-DGF patient and the value after dialysis finished for DGF patient. Denote the corresponding day  $d_0$ 

- 2. Find the time interval between  $d_0$  and 30 where  $Y_{1/2} < Y_i$  and  $Y_{1/2} > Y_{i+1}$ . If no such interval, then report "NA" for that patient.
- 3. The approximate ½ life time is  $d_{1/2} = \frac{Y_{1/2} Y_i}{Y_{i+1} Y_i} (d_{i+1} d_i) + d_i$

## 8.2. Safety Analyses

## 8.2.1. Overview of Planned Analyses

The safety analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 4 provides an overview of the planned analyses with further details of data displays being presented in Appendix 11.10: List of Data Displays.

 Table 4
 Overview of Planned Safety Analyses

| Endpoint / | | Abso | olute | | C | Change from Baseline | | |
|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | Summary | | Indiv | Individual | | Summary | | ridual |
| Type | T | F | F | L | T | F | F | L |
| Adverse Events <sup>1</sup> | | | | | | | | |
| All | Y | | | Y | | | | |
| Drug-Related | Y | | | Y | | | | |
| Serious | Y | | | Y | | | | |
| Leading to | Y | | | Y | | | | |
| Withdrawal | | | | | | | | |
| Laboratory Assessme | ents | | | | | | | |
| Haematology | Y | | | Y | | | | |
| Clinical Chemistry <sup>2</sup> : | Y | | | Y | | | | |
| Routine Urinalysis: | | | | Y | | | | |
| ECG | | | | | | | | |
| ECG Findings | Y | | | Y | | | | |
| ECG Measures | Y | | | Y | Y | Y | | Y |
| Vital Signs | Vital Signs | | | | | | | |
| Vital Signs | Y | | | Y | | Y | Y | |
| Immunogenicity | | | | | | | | |
| Frequency of Anti- | | | | Y | | | | |
| drug antibodies | | | | | | | | |
| ADA titers | | | | Y | | | | |

#### **NOTES:**

- T = Table, F = Figure, L = Listing, Y = Yes display generated..
- Summary represents any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual represents any displays of individual subject observed raw data.
- 1. Listings will include subject's numbers for individual AE's & AE system organ classes, preferred terms and verbatim text.

| Endpoint / | Absolute | | | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Parameter/ Display | Sum | mary | Indiv | ridual | Sum | mary | Individual | |
| Type | T | F | F | L | T | F | F | L |

Chemistry (includes LFTs and lipids) & haematology/coag summaries will include both changes from baseline & emergent results by PCI criteria. Listings for subjects with abnormalities of PCI will be prepared.

## 8.3. Pharmacokinetic Analyses

## 8.3.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

Table 5 provides an overview of the planned analyses with full details being presented in Appendix 11.10: List of Data Displays.

Table 5 Overview of Planned Pharmacokinetic Analyses

| Endpoints | Untransformed | | | | I | Log-Trai | nsforme | d |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | F | T | F | L | F | T | F | L |
| Plasma Drug Concentrations | $Y^{23}$ | $Y^3$ | $Y^1$ | Y | | | | |
| Derived PK Parameters | | $Y^3$ | | Y | | $Y^3$ | | |

#### **NOTES:**

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Mean (Linear and Semi-Log on same display) and Median (Linear and Semi-Log on same display) plots will be created.
- 3. Displays generated using the "PK" populations.

#### **8.3.2. Drug Concentration Measures**

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.2 Reporting Process & Standards).

#### **8.3.3.** Pharmacokinetic Parameters

#### **8.3.3.1.** Deriving Pharmacokinetic Parameters

• Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.2 Reporting Process & Standards).


GSK1070806

- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix Win Nonlin.
- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 6 will be determined from the plasma GSK1070806 concentration-time data, as data permits.
- Any deviation from the planned analyses will be described in detail in the study report.

Table 6 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve until the last time point of PK sample. Partial AUCs such as over 7, 30 or 90 days may be generated if deemed necessary. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Lamda_z | Terminal phase rate constant |
| | The number of points to determine Lambda_z |
| | The first point used to determine Lambda_z |
| | The last point used to determine Lambda_λz |
| t1/2 | Apparent terminal half-life will be calculated as: |
| | $t\frac{1}{2} = \ln 2 / Lambda_z$ |
| AUC(0-∞) | Area under the concentration time curve from predose to infinity. |

#### **NOTES:**

Additional parameters may be included as required.

## 9. OTHER STATISTICAL ANALYSES

# 9.1. Overview of Planned Pharmacokinetic / Pharmacodynamic Analyses

The pharmacokinetic / pharmacodynamic (PK/PD) analyses will be based on the "All Subjects" population, unless otherwise specified.

For the other biomarker variables/PD endpoints, summary tables will be reviewed to identify those biomarker variables/PD endpoints where there is a potential trend. If there is a trend then exploratory plots (scatter plots) will be presented for individual and/or pooled plasma GSK1070806 concentrations versus corresponding biomarker variables/PD endpoints (e.g. IL-18, IP-10).

 Table 7 provides an overview of the planned PK/PD analyses with further details of data displays being presented in Appendix 11.10: List of Data Displays. Any deviation from the planned analyses or additional analyses performed based on emerging data will be described in detail in the study report.

Table 7 Overview of Planned PK/PD Analyses

| Endpoints | Absolute | | | |
|---|---|---|---|---|
| | Sum | mary | Indiv | idual |
| | F | Т | F | L |
| Serum IL-18 (drug bound, total or free) vs. PK Plasma<br>Concentrations | Y | | | |


GSK1070806

| Endpoints | | Absolute | | |
|-----------|-----|----------|-------|--------|
| | Sum | mary | Indiv | ridual |
| | F | T | F | L |

## **NOTES:**

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 10. REFERENCES

GlaxoSmithKline Document Number 2015N240632\_01 : A Phase 2 Pilot, Single Arm Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of GSK 1070806 plus Standard of Care for the Prevention of Delayed Graft Function in Adult Subjects After Renal Transplantation Effective date: 03-FEB-2016

# 11. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4: | Analysis Populations |
| Section 11.1 | Appendix 1: Protocol Deviation Management and Definitions for Per<br>Protocol Population |
| | General Considerations for Data Analyses & Data Handling |
| Conventions | |
| Section 11.2 | Appendix 2: Time and Events |
| Section 11.3 | Appendix 3: Treatment States & Phases |
| Section 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 11.5 | Appendix 5: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| | Pharmacokinetic |
| | Pharmacodynamic / Biomarkers |
| Section 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| | Handling of Missing Dates |
| | Handling of Partial Dates |
| Section 11.7 | Appendix 7: Values of Potential Clinical Importance |
| | Laboratory Values |
| | • ECG's |
| | Vital Signs |
| Other RAP App | pendices |
| Section 11.88 | Appendix 8: Abbreviations & Trade Marks |
| Section 11.9 | Appendix 9: List of Data Displays |
| Section 11.10 | Appendix 10: Example Mock Shells for Data Displays |

# 11.1. Appendix 1: Protocol Deviation Definitions for Per Protocol Population

## 11.1.1. Exclusions from Per Protocol Population

A subject meeting any of the following criteria will be excluded from the Per Protocol population:

| Nun | nber | <b>Exclusion Description</b> |
|-----|------|--------------------------------------------------|
| 0 | )1 | Subject takes prohibited Concomitant Medications |
| 0 | )2 | Others as defined in the PDMP |

**NOTES:** For the details for prohibited concomitant medications, please refer to protocol Section 6.11.2

# 11.2. Appendix 2: Time and Events

| Study Day <sup>1</sup> | Screening | Pre-operative (baseline) | Intra-<br>operative (D0) | 4-8h <sup>2</sup> | D1 | D2 | Daily<br>until<br>discharge | Discharge | D30 | D90 | 6 & 12<br>months <sup>13</sup> | Unschedule<br>d Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed Consent/Demographics | X | | | | | | | | | | | |
| Medical/drug/alcohol/tobacco history | X | | | | | | | | | | | |
| GSK1070806 IV Infusion | | ← | • | | | | | | | | | |
| Kidney preservation fluid IL-18 | | | $X^{16}$ | | | | | | | | | |
| Kidney biopsy (post-reperfusion) <sup>3</sup> | | | X (~45 min) | | | | | | | | | |
| Clinical biopsy reports (if applicable) | | ← | | | | | | | | | | |
| Concomitant medication | X | X | X <sup>17</sup> | X | X | X | X | X | X | X | X | X |
| Evidence of infection | X | | | X | X | X | X | X | X | X | X | X |
| SAE / AE monitoring | ← | | | | | | | | | | | |
| DGF status (up to day 7) | | | | ← | | <del>-</del> | · | | | | | |
| Urine output | | X (native output) | X | X | X | X | X | X | | | | |
| Dialysis events since last assessment | | X | | X | X | X | X | X | X | X | X | X |
| Graft survival | | | ← | | | | | <del>-</del> | | | | |
| Viral serology (recipient & donor – HIV,<br>Hep B/C, EBV) <sup>4</sup> | X <sup>5</sup> | X | | | | | | | | | X | X |
| Viral serology (recipient & donor -herpes, varicella) <sup>4</sup> | | X | | | | | | | | | | |
| CMV monitoring | $X^5$ | X | | | | | | | | | X | X |
| BK virus monitoring <sup>6</sup> | | X | | | | | | | X | X | X | X |
| Vital signs <sup>7</sup> | X | | | X | X | X | X | X | X | X | X | X |
| Complete physical | X | | | | | | | | | | X | X |
| 12-lead ECG | X | | | | | | | X | | | X | X |
| Hematology / Clinical Chemistry /<br>Urinalysis | X | | | X | X | X | X | X | X | X | X | X |
| Pregnancy test <sup>8</sup> | X | | | | | | | | X | X | X | X |
| Serum cytokines / PD biomarkers | | X <sup>11</sup> | X (~45 min at biopsy) | X | X | X | | X | X | X | X | X |

| Study Day <sup>1</sup> | Screening | Pre-operative (baseline) | Intra-<br>operative (D0) | 4-8h <sup>2</sup> | D1 | D2 | Daily<br>until<br>discharge | Discharge | D30 | D90 | 6 & 12<br>months <sup>13</sup> | Unschedule<br>d Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Free, GSK1070806 bound & total IL18 9 | | $X^{11}$ | X (~45 min at biopsy) | X | X | X | | X | X | X | X | X |
| Pharmacokinetics <sup>9,10</sup> | | $X^{11}$ | X (~45 min at biopsy) | X | X | | | X (@168<br>hrs or at<br>earlier<br>discharge) | X | X | X | X |
| Immunogenicity 12 | | X <sup>11</sup> | | | | | | | X | X | X | X |
| Urinary biomarkers | | $X^{11}$ | | X | X | X | X | X | X | X | X | X |
| Peripheral blood leucocyte flow phenotyping 14 | | X | | | | | | X | | X | X | |
| PBMCs frozen for in vitro stimulation assays 14 | | X | | | | | | X | | X | X | |
| PBMCs placed in trizol for transcriptomic analysis <sup>14</sup> | | X | | | | | | X | | X | X | |

- 1. Day 0 defined as the calendar day of transplant.
- 2. Time post reperfusion.
- 3. Biopsies during transplantation may be 'core or wedge' at the discretion of the operating surgeon. If, in the judgement of the operating surgeon, biopsy poses unwarranted risk to the patient, it may be omitted.
- 4. Viral serology will include HIV, HBsAg, anti-HBs, anti-HBs antibodies, and hepatitis C antibody (if hepatitis C antibody positive, a hepatitis C RIBA immunoblot or polymerase chain reaction assay should be reflexively performed on the same sample to confirm the results as per NHS standard procedure), and serology for herpes simplex virus, Epstein Barr virus, and varicella zoster virus.
- 5. Screening viral status may be the most recent value recorded in the patient's medical records.
- 6. If BK positive then follow up screening should be implemented.
- 7. Vital signs will include systolic and diastolic blood pressure, pulse rate, and temperature.
- 8. Pregnancy testing will be performed in women of childbearing potential. Screening test may be urine or serum.
- 9. Sampling time points may be adjusted as appropriate based on emerging data.
- 10. PK sampling time points are as follows: predose, 45 min to 1 hr into infusion (coinciding with biopsy), 4-8 hrs, 24 hrs, 168 hrs (or pre-discharge if discharge before day 7), day 30 day 90, 6 and 12 months. Exact PK sampling time is to be recorded.
- 11. Blood and urine samples for immunogenicity and biomarker analyses must be collected prior to infusion with GSK1070806
- 12. For any non-completer a serum sample for immunogenicity testing will be taken 12 mths post-operatively.
- 13. For subjects who withdraw from study, where possible, assessments should continue according to the Time and Events table. The 6 and 12 mth safety follow-up should be performed.
- 14. Samples for subjects from Cambridge site only.
- 15. GSK1070806 can be infused any time during the pre-operative and/or intra-operative periods, but infusion <u>must</u> be complete prior to reperfusion of the allograft.


## GSK1070806

- 16. Sample to be obtained at time of back-table allograft preparation.17. Documentation of anaesthetics excluded.

## 11.3. Appendix 3: Treatment States and Phases

## 11.3.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment, unless otherwise specified.

| <b>Treatment Phase</b> | Definition |
|------------------------|---------------------------------------------|
| Pre-Treatment | Date/Time ≤ Study Treatment Start Date/Time |
| Post-Treatment | Date /Time> Study Treatment Stop Date/Time |

**Treatment Description** 

| Code | Treatment Description | Final Data Display (i.e. HARP/other) |
|------|-----------------------|--------------------------------------|
| A | 3 mg/kg GSK1070806 | 3 mg/kg GSK1070806 |

#### 11.3.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date/time of the study treatment.

## 11.3.3. Treatment States for AE Data

| <b>Treatment State</b> | Definition |
|---|---|
| AE = Pre-<br>Treatment | AE Start Date/Time < Study Treatment Start Date/Time |
| AE Onset Time | If Treatment Start Date/Time > AE Onset Date/Time : |
| Since 1st Dose | = AE Onset Date - Treatment Start Date |
| (Days) | If Treatment Start Date ≤ AE Onset Date : |
| | = AE Onset Date – Treatment Start Date + 1 |
| | Missing otherwise |
| AE Duration<br>(Days) | AE Resolution Date/Time – AE Onset Date/Time (follow SOP) |
| AE = Drug-related | If relationship is marked 'YES' on [Inform/CRF OR value is missing. |

#### **NOTES:**

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment

## 11.4. Appendix 4: Data Display Standards & Handling Conventions

#### 11.4.1. Baseline Definition & Derivations

#### 11.4.1.1. Baseline Definitions

For all endpoints baseline value will be the latest pre-dose assessment.

## 11.4.1.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Baseline Visit Value – Baseline |
| [% Change from Baseline] | = [ (Post-Baseline Visit Value – Baseline) / Baseline ] x 100] |

#### NOTE:

- Unless otherwise specified, the baseline definitions specified in 11.4.1.1Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 11.4.2. Reporting Process & Standards

| <b>Reporting Process</b> | Reporting Process |
|---|---|
| Software | |
| <i>y</i> . | pported versions of SAS and R software will be used to perform all merate tables, figures, and listings. |
| Reporting Area | |
| HARP Server | : <u>Us1salx00259-HARP PROD-US</u> |
| HARP Area | : \ARPROD\GSK1070806\204882 |
| QC Spreadsheet | QC Spreadsheet :\ARWORK\GSK1070806\204882\ReportingEffort\Documents |
| <b>Analysis Datasets</b> | Analysis Datasets |
| <ul> <li>Analysis datasets will be created according to Integrated Data Standards Library<br/>standards.</li> </ul> | |
| Generation of RTF I | Files |
| RTF files will be | generated for SAC tables. |

## **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings

- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- In the top left header on each page of output the study part will be indicated after the protocol number (ie, "204824")
- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
- Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables or figures, unless otherwise stated.
- All unscheduled visits will be listed.

| D | • | 4 • | • | 04 4. 4. |
|---------------------------|------|------|---------|-------------------|
| 1100 | crin | TIVE | Summary | <b>Statistics</b> |
| $\mathbf{p}_{\mathbf{c}}$ | CLID | 4 | Summar | Dualistics |

| 1 | <b>V</b> |
|------------------|--------------------------------------------|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |

## **Reporting of Pharmacokinetic Concentration**

| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
|---|---|
| Summary Statistics | Handling NQ values per GUI_51487 |
| Reporting of Pharm | nacokinetic Parameters |
| Descriptive | N, n, geometric mean, 95% CI of geometric mean, standard |
| Summary Statistics | deviation (SD) of logged data and between geometric coefficient of |
| (Log Transformed | variation ( $CV_{b/w}$ (%)): |
| Data) | $CV_b$ (%) = $\sqrt{(\exp(SD^2) - 1) * 100}$ |
| | (NOTE: SD is the SD of log transformed data) |
| Parameters Not | tmax, first point, last point and number of points used in the |
| Being Log | determination of Lambda_λz. |
| Transformed | |
| Parameters Not | tmax, first point, last point and number of points used in the |
| Being Summarised | determination of Lambda_λz. |
| Listings | Include the first point, last point and number of points used in the |
| | determination of Lambda_λz. |
| Cranbinal Displays | |

## **Graphical Displays**

- Refer to IDSL Statistical Principles 7.01 to 7.13.
- The same symbol and line type will be used across figures to represent a given treatment group.
- X-axis variables of time and dose will be plotted as continuous numeric variables.

## 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

## **Study Day**

- Calculated as the number of days from dosing date :
  - [1] Assessment Date = Missing  $\rightarrow$  Study Day = Missing
  - [2] Assessment Date < Transplant Date → Study Day = Assessment Date Transplant Date
  - [3] Assessment Data ≥ Transplant Date → Study Day = Assessment Date Transplant Date

## 11.5.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - [1] Any subject with a missing day will have this imputed as day '15'.
  - [2] Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

## 11.5.3. Safety

#### +++ ECG Parameters +++

#### **RR** Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as:
  - o If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

o If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

• If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

## Corrected QT Intervals

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTCF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

## +++ Laboratory Parameters +++

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x ' becomes x 0.01
  - Example 2: 1 Significant Digit = > x' becomes x + 0.1
  - Example 3: 0 Significant Digits = < x' becomes x 1.
- If there is more than one value of a particular parameter for a subject for a visit, the scheduled value will be used in summary; all values will be listed.

#### 11.5.4. Pharmacokinetic

#### **GSK1070806 Derived PK Parameters**

• Refer to PK Guidance document GUI00000051487: Non-compartmental Analysis of Pharmacokinetic Data for more information.

# 11.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

## 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion was defined as Safety who either prematurely withdrawn or completed FU visits and assessments. |
| | Withdrawn subjects were not replaced in the study. |
| | All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |

# 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | • Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul><li>[1] These data will be indicated by the use of a "blank" in subject listing displays.</li><li>[2] Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li></ul> |
| Outliers | • Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |
| Biomarkers<br>Free IL-18<br>Drug<br>Bound IL-<br>18 and<br>total IL-18 | • LLQ will be set as LLQ/2 |
| | • ULQ will be set as ULQ |
| | <ul> <li>Values used for the computation of the change from baseline and for<br/>summaries, plots and analysis, if deemed applicable.</li> </ul> |
| | • Number of data imputed will be highlighted in the summaries where as listings will report the values as below LLQ or above ULQ. |
| | • If more than a third of obs are below LLQ or above LLQ then no imputation will be performed for that subject. |
| | • To enable the data to be plotted (i.e. some groups may remain below BLQ) this rule may not be applied to Free & Drug Bound IL18 parameters. |

## 11.6.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | • The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be |

| Element | Reporting Detail |
|---|---|
| | applied for calculating the time to onset and the duration of the event: |
| | <ul> <li>For a missing start day, the 1st of the month will be used unless this is before the start date of investigational product; in this case the study treatment start date will be used (and hence the event is considered On-treatment as per Section 11.3: Treatment States and Phases.</li> <li>For a missing stop day, the last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |
| | • Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied. |

# 11.6.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | • Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | • Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |


GSK1070806

# 11.6.2.3. Handling of Missing Data for Statistical Analysis/Efficacy Endpoints

| Element | Reporting Detail |
|-----------|-------------------------------------|
| All | Missing values will not be imputed. |
| Endpoints | |
# 11.7. Appendix 7: Values of Potential Clinical Importance

## 11.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | Δ from<br>BL | ↓0.075 | |
| | | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | Δ from<br>BL | ↓25 | |
| Lymphocytes | GI/L | | 0.8 | |
| Neutrophil Count | GI/L | | 1.5 | |
| Platelet Count | GI/L | | 100 | 550 |
| While Blood Cell Count (WBC) | GI/L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| <b>Laboratory Parameter</b> | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | G/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | Δ from<br>BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Magnesium | mmol/L | | 0.5 | 1.23 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | IU/L | High | ≥ 2x ULN |
| AST/SGOT | IU/L | High | ≥ 2x ULN |
| AlkPhos | IU/L | High | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | μmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

## 11.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|-------------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | > 450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 110 |
| Change from Baseline | | | |
| Increase from Baseline<br>QTc | msec | > 60 | |

## 11.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |
| Temperature | °C | 35.5 | 37.5 |

# 11.8. Appendix 8 – Abbreviations & Trade Marks

## 11.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| AE | Adverse Event |
| GSK | GlaxoSmithKline |
| ADA | Anti-Drug Antibodies |
| AUC | Area under concentration-time curve |
| AUC(0-∞) | Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time |
| BMI | Body mass index |
| BPM | Beat Per Minute |
| CL | Systemic clearance of parent drug |
| Cmax | Maximum observed concentration |
| CI | Confidence Interval |
| CV | Coefficient of variance |
| HR | Heart rate |
| ICH | International Conference on Harmonization of Technical Requirements |
| | for Registration of Pharmaceuticals for Human Use |
| IDSL | Integrated Data Standards Library |
| Kg | Kilogram |
| $\lambda z$ | Terminal phase rate constant |
| LLQ | Lower limit of quantification |
| NQ | Non-quantifiable concentration measured as below LLQ |
| PK | Pharmacokinetic |
| QC | Quality control |
| RAP | Reporting and Analysis Plan |
| SAS | Statistical Analysis Software |
| SI | System Independent |
| SD | Standard deviation |
| SOP | Standard Operating Procedure |
| t OR tlast | Time of last observed quantifiable concentration |
| t½ | Terminal phase half-life |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| tmax | Time of occurrence of Cmax |
| ULQ | Upper limit of quantification |
| ULN | Upper limit of normal |
| UK | United Kingdom |

## 11.8.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies | Trademarks not owned by the GlaxoSmithKline Group of Companies |
|---|---|
| NONE | NONMEM |
| | SAS |
| | WinNonlin |

# 11.9. Appendix 9: List of Data Displays

## 11.9.1. Deliverable

| Delivery | Description |
|---|---|
| IA1 | Interim analysis after recruitment of approximately 8 to 10 patients to review for a consideration of dose adjustment |
| IA2 | Interim analysis once the last patient completes 7-Days post-transplant. |
| SAC | Final Statistical Analysis Complete |

## 11.9.2. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|--------------|--------------|
| Study Population | 1.01 to 1.10 | N/A |
| Efficacy | 2.01 to 2.29 | 2.01 to 2.17 |
| Safety | 3.01 to 3.24 | N/A |
| Pharmacokinetic | 4.01 to 4.03 | 4.01 to 4.03 |
| PK/PD | NA | 5.01 |
| Section | Listings | |
| ICH Listings | 1 to 19 | |
| Other Listings | 20 to 41 | |

# 11.9.3. Study Population Tables

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable |
| Subject | Disposition | | | | |
| 1.01 | All<br>Subjects | ES1 | Summary of Subject Disposition | | IA2, SAC |
| 1.02 | All<br>Subjects | ES6 | Summary of Reasons for Screening Failure | | IA2, SAC |
| 1.03 | All<br>Subjects | DV1a | Summary of Important Protocol Deviations | | IA2, SAC |
| 1.04 | All<br>Subjects | SA2 | Summary of Deviations Leading to Exclusion from Per Protocol Population | | IA2, SAC |
| 1.05 | All<br>Subjects | ES5 | Summary of Reasons for Withdrawals | | IA2, SAC |
| Demogr | raphics | | | | |
| 1.06 | All<br>Subjects | DM1 | Summary of Demographic Characteristics | | IA2, SAC |
| 1.07 | All<br>Subjects | DM5 | Summary of Race and Racial Combinations | | IA2, SAC |
| 1.08 | All<br>Subjects | SA1 | Summary of Study Populations | | IA2, SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable |
| Medica | Medical Condition & Con Meds | | | | |
| 1.09 | All<br>Subjects | MH1 | Summary of [Current/Past] Medical Conditions | | IA2, SAC |
| 1.10 | All<br>Subjects | CM1 | Summary of Most Frequently used<br>Concomitant Medications by Generic Term | Footnote: Most Frequently means the overall concomitant medication used is >= 10% | IA1, IA2,<br>SAC |

# 11.9.4. Efficacy Tables

| Effica | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| DGF | | | | | |
| 2.01 | Analysis<br>Population | Non-Standard<br>EFF_T3 | Proportion of Subjects with DGF | | IA1, IA2,<br>SAC |
| 2.02 | Per<br>Protocol | Non-Standard<br>EFF_T3 | Proportion of Subjects with DGF | | IA2, SAC |
| Graft | function | | | | |
| 2.03 | Analysis<br>Population | Non-Standard<br>EFF_T1 | Summary Statistics of Serum Creatinine | | IA1, IA2,<br>SAC |
| 2.04 | Analysis<br>Population | Non-Standard<br>EFF_T2 | Summary of Serum Creatinine Change from Baseline | | IA1, IA2,<br>SAC |
| 2.05 | Analysis<br>Population | Non-Standard<br>EFF_T1 | Summary Statistics of AUC of 7 Day Serum<br>Creatinine | Only consider patients who have Day 7 serum creatinine value | IA1, IA2,<br>SAC |
| 2.06 | Analysis<br>Population | Non-Standard<br>EFF_T1 | Summary Statistics of AUC of 30 Day Serum Creatinine | | IA1, IA2,<br>SAC |
| 2.07 | Analysis<br>Population | Non-Standard<br>EFF_T1 | Summary Statistics of ½ -Life of 30 Day Serum Creatinine | | IA1, IA2,<br>SAC |

| Effica | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 2.08 | All<br>Subjects | Non-Standard<br>EFF_T4 | Proportion of Subjects with Renal Functional<br>Graft within 7 Days after Transplant | Including primary non function;3 day functional DGF; 7 day functional DGF; 3 day intermediate graft function; 7 day intermediate graft function; 3 day immediate graft function; 7 day immediate graft function | IA1, IA2,<br>SAC |
| Acute | rejection ris | k | | | |
| 2.09 | All<br>Subjects | Non-Standard<br>EFF_T3 | Proportion of Subjects with Episodes of Biopsy-<br>Proven Acute Rejection | | IA2, SAC |
| 2.10 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of Episodes of Biopsy-<br>Proven Acute Rejection | | IA2, SAC |
| PD bio | marker | ı | | | |
| 2.11 | All<br>Subjects | Non-Standard<br>EFF_T1 | Summary Statistics of Serum IP-10 | | IA2, SAC |
| 2.12 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of Serum IP-10 Change from Baseline | | IA2, SAC |
| 2.13 | All<br>Subjects | Non-Standard<br>EFF_T1 | Summary Statistics of Mig | | IA2, SAC |
| 2.14 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of Mig Change from Baseline | | IA2, SAC |

| Effica | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 2.15 | All<br>Subjects | Non-Standard<br>EFF_T1 | Summary Statistics of Free IL-18 | | IA2, SAC |
| 2.16 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of Free IL-18 Change from Baseline | | IA2, SAC |
| 2.17 | All<br>Subjects | Non-Standard<br>EFF_T1 | Summary Statistics of Bound IL-18 | | IA2, SAC |
| 2.18 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of Bound IL-18 Change from Baseline | | IA2, SAC |
| 2.19 | All<br>Subjects | Non-Standard<br>EFF_T1 | Summary Statistics of Total IL-18 | | IA2, SAC |
| 2.20 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of total IL-18 Change from Baseline | | IA2, SAC |
| Urine | biomarker | | | | |
| 2.21 | All<br>Subjects | Non-Standard<br>EFF_T1 | Summary Statistics of IL-18 | | IA2, SAC |
| 2.22 | All<br>Subjects | Non-Standard<br>EFF_T1 | Summary Statistics of NGAL | | IA2, SAC |
| 2.23 | All<br>Subjects | Non-Standard<br>EFF_T1 | Summary Statistics of KIM1 | | IA2. SAC |

| Effica | Efficacy Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| Dialys | is dependenc | y and graft surv | rival | | |
| 2.24 | All<br>Subjects | Non-Standard<br>EFF_T3 | Proportion of Subjects Who are Dialysis-<br>Independent at Visits up to 12 Months post<br>Transplant | | IA2, SAC |
| Exploi | ratory | , | | | |
| 2.25 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of % Free GSK1070806 within Renal Graft Biopsies | | IA2, SAC |
| 2.26 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of % Bound GSK1070806 within Renal Graft Biopsies | | IA2, SAC |
| 2.27 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of Level of IL-18 in Renal Preservation Fluid | | IA2, SAC |
| 2.28 | All<br>Subjects | Non-Standard<br>EFF_T2 | Summary Statistics of Serum Cytokine Levels | | IA2, SAC |
| 2.29 | All<br>Subjects | Non-Standard<br>EFF_T1 | Summary Statistics of Length of Hospital Stay | | IA2, SAC |

# 11.9.5. Efficacy Figures

| Effica | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| Serum | Creatinine | | | | |
| 2.01 | All<br>Subjects | Non-Standard<br>EFF_F1 | Individual Line Plot of Serum Creatinine over Time | Including the mean line plot; starting from baseline | IA1, IA2,<br>SAC |
| 2.02 | All<br>Subjects | Non-Standard<br>EFF_F1 | Individual Line Plot of Serum Creatinine<br>Change from Baseline over Time | Including the mean line plot | IA1, IA2,<br>SAC |
| Graft | function | | | | |
| 2.03 | All<br>Subjects | Non-Standard<br>EFF_F2 | Individual Line Plot of Urine Output over Time | | IA2, SAC |
| 2.04 | All<br>Subjects | Non-Standard<br>EFF_F3 | Kaplan-Meier Curve of Graft Survival up to 12<br>Months post Transplant | | IA2, SAC |
| PD bio | markers | | | | |
| 2.05 | All<br>Subjects | Non-Standard<br>EFF_F1 | Individual Line Plot of Serum IP-10 over Time | Including the mean line plot; starting from baseline | IA2, SAC |
| 2.06 | All<br>Subjects | Non-Standard<br>EFF_F1 | Individual Line Plot of Serum IP-10 Change from Baseline over Time | Including the mean line plot | IA2, SAC |
| 2.07 | All<br>Subjects | Non-Standard<br>EFF_F1 | Individual Line Plot of Serum Mig over Time | Including the mean line plot; starting from baseline | IA2, SAC |

| Effica | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 2.08 | All<br>Subjects | Non-Standard<br>EFF_F1 | Individual Line Plot of Serum Mig Change from Baseline over Time | Including the mean line plot | IA2, SAC |
| 2.09 | All<br>Subjects | Non-Standard<br>EFF_F1 | Individual Line Plot of Serum IL-18 Levels over Time | Including free IL-18; bound IL-18 and total IL-18 Including the mean line plot | IA1, IA2,<br>SAC |
| 2.10 | All<br>Subjects | Non-Standard<br>EFF_F1 | Individual Line Plot of Serum IL-18 Levels<br>Change from Baseline over Time | Including free IL-18; bound IL-18 and total IL-18 Including the mean line plot | IA2, SAC |
| Urine | Biomarkers | | | | |
| 2.11 | All<br>Subjects | Non-Standard<br>EFF_F3 | Mean (95% CI) Plot of Urine IL-18 | Two sided confidence interval | IA2, SAC |
| 2.12 | All<br>Subjects | Non-Standard<br>EFF_F3 | Mean (95% CI) Plot of Urine NGAL | Two sided confidence interval | IA2, SAC |
| 2.13 | All<br>Subjects | Non-Standard<br>EFF_F3 | Mean (95% CI) Plot of Urine KIM1 | Two sided confidence interval | IA2, SAC |
| Exploi | Exploratory | | | | |
| 2.14 | All<br>Subjects | Non-Standard<br>EFF_F2 | Individual Line Plot of Serum IL-18 Binding<br>Protein over Time | starting from baseline | IA2, SAC |
| 2.15 | All<br>Subjects | Non-Standard<br>EFF_F2 | Individual Line Plot of Serum Cytokine Levels over Time | starting from baseline | IA2, SAC |

| Efficacy Figures | | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 2.16 | All<br>Subjects | Non-Standard<br>EFF_F1 | Individual Line Plot of Serum Cytokine Levels<br>Change from Baseline over Time | Including the mean line plot | IA2, SAC |
| Patien | Patient Profile | | | | |
| 2.17 | All<br>Subjects | Non-Standard<br>EFF_F5 | Patient Profile Plot of Biomarker/PD Endpoints | Incuding serum IP-10; serum mig; free IL-18; bound IL-18; total IL-18 | IA2, SAC |

# 11.9.6. Safety Tables

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| Adver | se Events – ( | Overall | | | |
| 3.01 | All<br>Subjects | AE1 | Summary of All Adverse Events | | IA1, IA2,<br>SAC |
| 3.02 | All<br>Subjects | AE3 | Summary of Common Adverse Events by<br>Preferred Term | Common AE = Frequency > 1% | IA1, IA2,<br>SAC |
| 3.03 | All<br>Subjects | AE1 | Summary of Drug-Related Adverse Events by<br>System Organ Class | | IA1, IA2,<br>SAC |
| 3.04 | All<br>Subjects | AE1 | Summary of Serious Adverse Events by System<br>Organ Class | | IA1, IA2,<br>SAC |
| 3.05 | All<br>Subjects | AE1 | Summary of Adverse Events Leading to<br>Withdrawals from Study or Study Treatment | | IA1, IA2,<br>SAC |
| Adver | se Events – i | n patients (befor | re discharge) | | |
| 3.06 | All<br>Subjects | AE1 | Summary of All Adverse Events before Discharge | | IA2, SAC |
| 3.07 | All<br>Subjects | AE3 | Summary of Common Adverse Events by<br>Overall Frequency before Discharge | | IA2, SAC |
| 3.08 | All<br>Subjects | AE5 | Summary of Drug-Related Adverse Events by<br>System Organ Class before Discharge | | IA2, SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.09 | All<br>Subjects | AE1 | Summary of Serious Adverse Events by System<br>Organ Class before Discharge | | IA2, SAC |
| 3.10 | All<br>Subjects | AE1 | Summary of Adverse Events Leading to<br>Withdrawals from Study / Permanent<br>Discontinuation of Study Treatment before<br>Discharge | | IA2, SAC |
| Adver | se Events – o | ut patients (afte | r discharge) | | |
| 3.11 | All<br>Subjects | AE1 | Summary of All Adverse Events after Discharge | | IA2, SAC |
| 3.12 | All<br>Subjects | AE3 | Summary of Common Adverse Events by<br>Overall Frequency after Discharge | | IA2, SAC |
| 3.13 | All<br>Subjects | AE5 | Summary of Drug-Related Adverse Events by<br>System Organ Class after Discharge | | IA2, SAC |
| 3.14 | All<br>Subjects | AE1 | Summary of Serious Adverse Events by System<br>Organ Class after Discharge | | IA2, SAC |
| 3.15 | All<br>Subjects | AE1 | Summary of Adverse Events Leading to<br>Withdrawals from Study / Permanent<br>Discontinuation of Study Treatment after<br>Discharge | | IA2, SAC |
| Labs | Labs | | | | |
| 3.16 | All<br>Subjects | LB1 | Summary of Chemistry Changes from Baseline | | IA2, SAC |

| Safety | Safety Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 3.17 | All<br>Subjects | LB1 | Summary of Emergent Chemistry Results of Potential Clinical Importance | | IA1, IA2,<br>SAC |
| 3.18 | All<br>Subjects | LB1 | Summary of Haematology Changes from Baseline | | IA2, SAC |
| 3.19 | All<br>Subjects | LB1 | Summary of Emergent Haematology of Potential Clinical Importance | | IA1, IA2,<br>SAC |
| Vital S | Signs | | | | |
| 3.20 | All<br>Subjects | VS1 | Summary of Change from Baseline in Vital Signs | Include the Respiration Rate and Temperature | IA2, SAC |
| 3.21 | All<br>Subjects | VS2 | Summary of Emergent Vital Signs Results of<br>Potential Clinical Importance | | IA1, IA2,<br>SAC |
| ECGs | | | | | |
| 3.22 | All<br>Subjects | EG1 | Summary of ECG Findings | | IA2, SAC |
| 3.23 | All<br>Subjects | Non-Standard<br>EFF_T5 | Frequency of Maximum Emergent QTc Values by Category | | IA1, IA2,<br>SAC |
| 3.24 | All<br>Subjects | EG2 | Summary of Change from Baseline in ECG<br>Values | | IA2, SAC |

## 11.9.7. Pharmacokinetic Tables

| Pharm | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK Co | ncentration | Data | | | |
| 4.01 | PK | PK01 | Summary of Plasma GSK1070806 Pharmacokinetic Concentration-Time Data (mg/mL) | | IA1, IA2,<br>SAC |
| PK De | rived Param | eters | | | |
| 4.02 | PK | PKPT1 | Summary Statistics of Derived Plasma<br>GSK1070806 Pharmacokinetic Parameters | Parameters with units | IA1, IA2,<br>SAC |
| 4.03 | PK | PKPT3 | Summary Statistics of Log-Transformed Derived Plasma GSK1070806 Pharmacokinetic Parameters | Parameters with units; exclude non-continuous PK parameters; | IA2, SAC |

# 11.9.8. Pharmacokinetic Figures

| Pharm | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| Indivi | dual Plots | | | | |
| 4.01 | PK | PKCF1P | Individual GSK1070806 Plasma Concentration-<br>Time Plot by Subject (Linear and Semi-Log) | Paginate by Subject | IA2, SAC |
| Mean | / Median Plo | ts | | | |
| 4.02 | PK | PKCF2 | Mean and Median Plasma GSK1070806<br>Concentration-Time Plots by Treatment (Linear and Semi-log) | | IA2, SAC |
| 4.03 | PK | PKCF3 | Median and Median Plasma GSK1070806<br>Concentration-Time Plots by Treatment (Linear<br>and Semi-log) | | IA2, SAC |

# 11.9.9. Pharmacokinetic / Pharmacodynamic Figures

| Pharm | Pharmacodynamic / Biomarker Figures | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 5.01 | PK | Non-Standard<br>PKPD_F1 | Scatter Plot of Free and Drug Bound IL-18<br>Serum Levels Versus GSK1070806 Plasma<br>Concentration | Panel: by free and drug bound IL-18 X-Axis: Plasma Concentration Y-Axis: free and drug bound IL-18 Add Footnote X-Axis: Untransformed data presented using Log10 scale | IA2, SAC |

# 11.9.10. ICH Listings

| ICH L | Listings | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| Subjec | ct Disposition | <u> </u> | | | |
| 1 | All<br>Subjects | ES2 | Listing of Reasons for Study Withdrawal | | IA1, IA2,<br>SAC |
| 2 | All<br>Subjects | ES7 | Listing of Reasons for Screening Failure | | IA1, IA2,<br>SAC |
| 3 | All<br>Subjects | SA3a | Listing of Subjects Excluded from Any Populations | | IA2, SAC |
| 4 | All<br>Subjects | DV2 | Listing of Important Protocol Deviations | | IA1, IA2,<br>SAC |
| 5 | All<br>Subjects | IE3 | Listing of Subjects with Inclusion/Exclusion<br>Criteria Deviations | | IA1, IA2,<br>SAC |
| Demog | graphics | | | | |
| 6 | All<br>Subjects | DM2 | Listing of Demographic Characteristics | | IA1, IA2,<br>SAC |
| 7 | All<br>Subjects | DM9 | Listing of Race | | IA1, IA2,<br>SAC |
| Expos | ure | | | | |

| ICH L | istings | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 8 | All<br>Subjects | EX3 | Listing of Exposure | | SAC |
| Adver | se Events | | | | |
| 9 | All<br>Subjects | AE7 | Listings of Subject Numbers for Individual<br>Adverse Events | | IA1, IA2,<br>SAC |
| 10 | All<br>Subjects | AE8 | Listing of All Adverse Events | | IA1, IA2,<br>SAC |
| 11 | All<br>Subjects | AE8 | Listing of Serious Adverse Events | | IA1, IA2,<br>SAC |
| 12 | All<br>Subjects | AE8 | Listing of Adverse Events Leading to<br>Withdrawal from Study | | IA1, IA2,<br>SAC |
| LABS | | | | | |
| 13 | All<br>Subjects | LB5 | Listing of Haematology Laboratory Data for<br>Subjects with Abnormalities of Potential<br>Clinical Importance | | IA1, IA2,<br>SAC |
| 14 | All<br>Subjects | LB5 | Listing of Clinical Chemistry Laboratory Data for Subjects Abnormalities of Potential Clinical Importance. | | IA1, IA2,<br>SAC |
| 15 | All<br>Subjects | UR2b | Listing of Urinalysis Data | | IA2, SAC |

| ICH L | istings | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | ID / Example Title | | Programming Notes | Deliverable |
| 16 | All<br>Subjects | Non-Standard<br>SAFE_L1 | Listing of Clinical Chemistry Laboratory Values (Total cholesterol, HDL, LDL, Triglycerides, Creatinine Clearance (MDRD) and Associated Ratios). | | IA2, SAC |
| ECGs | | | | | |
| 17 | All<br>Subjects | EG3 | Listing of ECG Values for Subjects with Abnormalities of Potential Clinical Importance. | | IA1, IA2,<br>SAC |
| Vital S | Signs | | | | |
| 18 | All<br>Subjects | CP_VS4 | Listing of Vital Signs for Subjects with<br>Abnormalities of Potential Clinical Importance | | IA1, IA2,<br>SAC |
| Immunogenicity | | | | | |
| 19 | All<br>Subjects | IMM2 | Listing of Immunogenicity Results | ADA tiers | IA2, SAC |

# 11.9.11. Non-ICH Listings

| Non-I | CH Listings | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK | | | | | |
| 20 | PK | PKCL1P | Listing of Plasma GSK1070806 Pharmacokinetic Concentration-Time Data | | IA2, SAC |
| 21 | PK | PKPL1P | Listing of Derived Plasma GSK1070806<br>Pharmacokinetic Parameters | Include dose and dose number | IA2, SAC |
| Graft | Function | | | | |
| 22 | Analysis<br>Population | Non-Standard SAFE_L1 | Listing of Individual Serum Creatinine | | IA1, IA2,<br>SAC |
| 23 | Analysis<br>Population | Non-Standard<br>SAFE_L1 | Listing of Individual AUC of 7 Day Serum<br>Creatinine | No change from baseline column | IA1, IA2,<br>SAC |
| 24 | Analysis<br>Population | Non-Standard<br>SAFE_L1 | Listing of Individual AUC of 30 Day Serum<br>Creatinine | No change from baseline column | IA1, IA2,<br>SAC |
| 25 | All<br>Subjects | Non-Standard<br>SAFE_L2 | Listing of Individual Graft Function in the First 7<br>Days | Including primary non function;3 day functional DGF; 7 day functional DGF; 3 day intermediate graft function; 7 day intermediate graft function; 3 day immediate graft function; 7 day immediate graft function | IA1, IA2,<br>SAC |

| Non-IO | CH Listings | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| 26 | All<br>Subjects | Non-Standard<br>SAFE_L2 | Listing of Individual Urine Output | Including change from baseline | IA2, SAC |
| 27 | All<br>Subjects | Non-Standard SAFE_L1 | Listing of Individual with Episodes of Biopsy-<br>Proven Acute Rejection | | IA2, SAC |
| Pharm | acodynamic | & Biomarkers | | | |
| 28 | All<br>Subjects | Non-Standard<br>EFF_L1 | Listing of Individual of IL-18 | | IA1, IA2,<br>SAC |
| 29 | All<br>Subjects | Non-Standard<br>EFF_L1 | Listing of Individual of NGAL | | IA2, SAC |
| 30 | All<br>Subjects | Non-Standard<br>EFF_L1 | Listing of Individual of KIM1 | | IA2, SAC |
| 31 | All<br>Subjects | Non-Standard<br>PD_L1 | Listing of Biomarkers | | IA2, SAC |
| 32 | All<br>Subjects | Non-Standard<br>PD_L1 | Listing of Free and Drug-bound IL-18 Levels In Serum | | IA2, SAC |
| Dialys | is dependenc | y and graft surv | ival | | |
| 33 | All<br>Subjects | Non-Standard<br>SAFE_L1 | Listing of Number of Dialysis Events per Patient in the First 30 Days Post Transplant | | IA1, IA2,<br>SAC |

| Non-I | CH Listings | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| Recipi | ent Kidney I | <b>Data</b> | | | |
| 34 | All<br>Subjects | Non-Standard SAFE_L3 | Listing of Recipient Virology | | IA2, SAC |
| Explo | ratory | | | | |
| 35 | All<br>Subjects | Non-Standard<br>SAFE_L1 | Listing of Individual % bound GSK1070806 within Renal Graft Biopsies | | IA2, SAC |
| 36 | All<br>Subjects | Non-Standard<br>SAFE_L1 | Listing of Individual Level of IL-18 in Renal<br>Preservation Fluid | | IA2, SAC |
| 37 | All<br>Subjects | Non-Standard<br>SAFE_L1 | Listing of Individual Change from Baseline<br>Histological Analysis of Biopsies with Respect<br>to Cellular Infiltrate | | IA2, SAC |
| 38 | All<br>Subjects | Non-Standard<br>SAFE_L2 | Listing of Individual of Length of Hospital and Re-hospitalization Stay | | IA1, IA2,<br>SAC |
| Donor | Kidney Data | a | | | |
| 39 | All<br>Subjects | Non-Standard<br>SAFE_L3 | Listing of Donor Virology | | IA2, SAC |
| 40 | All<br>Subjects | Non-Standard<br>SAFE_L4 | Listing of Donor Characteristics | Cold ischiemic time; warm ischemic time; age; sex; last creatinine before transplant; medical conditions; biopsy performed yes/no, transport system (ice or perfusion) | IA1, IA2,<br>SAC |

| Non-IO | Non-ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Populatio<br>n | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable |
| PK/PE | ) | | | | |
| 41 | PK | Non-Standard<br>SAFE_L5 | Listing of Serum IL-18 (drug bound, total or free) vs. PK Plasma Concentrations | | IA2, SAC |

11.10. Appendix 10: Example Mock Shells for Data Displays

204824

Example : EFF\_F1 Page 1 of X

Protocol : 204824
Population : All Subjects

Figure X Individual Subject Spaghetti Plot with Mean Line

NOTE: This is example only. Plot adjusted accordingly to study data.

204824

Example : EFF\_F2
Protocol : 204824


Population : All Subjects

Figure X Individual Subject Spaghetti Plot

NOTE: This is example only. Plot adjusted accordingly to study data.

204824

Example : EFF\_F3
Protocol : 204824


Population : All Subjects

Figure X Mean Plot of xxx

NOTE: Plot adjusted accordingly to study data


Example : EFF\_F4
Protocol : 204824
Population : All Subjects

Figure X
Kaplan-Meier Curve of Graft Survival up to 12 Months post Transplant



NOTE: Plot adjusted accordingly to study data, with plot also including the other treatments groups on subsequent pages.

Example : EFF\_F5 Page 1 of X

Protocol : 204824 Population : Safety

Figure X
Patient Profile Plot



NOTE: Plot adjusted accordingly to study data, with plot also including the other treatments group and parameters on subsequent pages.

Example : PKPD\_F1 Page 1 of X

Protocol : 204824 Population : All Subjects

Figure X
Scatter Plot of Free and Drug Bound IL-18 Serum Levels Versus GSK1070806 Plasma Concentration



Note: IL-18 Serum values defined as BLQ, are imputed as half of LLQ.

Note: Analysis numeric results in std units (NQ values not imputed with 0) are considered as Plasma Concentration values.

Note: Free IL-18 plot is not presented as majority of data is BLQ.

Note: Doses = 0.008. 0.05, 0.25, 1.0, 3.0 & 10 mg/kg HV

204824

Example : EFF\_T1 : 204824 Page 1 of X

Protocol Population : All Subjects

Table X Summary Statistics of XXX (unit)

**Summary: Absolute** 

| Treatment | N | Visit | Planned<br>Relevant<br>Time | n | Mean | S.D | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|
| GSK1070806 3 mg/kg | XX | XX | x | | xxx.x | XX.XX | xxx.x | XXX | XXX |
| | XX | | x | | xxx.x | XX.XX | XXX.X | XXX | XXX |
| | XX | XX | X | | XXX.X | XX.XX | XXX.X | XXX | XXX |
| | XX | | x | | XXX.X | XX.XX | XXX.X | XXX | XXX |

204824


Example : EFF\_T2 Protocol : 204824

Population : All Subjects

Table X
Summary Statistics of XXX (unit)

**Summary: Change from Baseline** 

| Treatment | N | Visit | Planned<br>Relevant<br>Time | n | Mean | S.D | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|
| GSK1070806 3 mg/kg | XX | XX | X | | XXX.X | XX.XX | XXX.X | XXX | xxx |
| | XX | | X | | XXX.X | xx.xx | XXX.X | xxx | XXX |
| | XX | XX | X | | XXX.X | XX.XX | XXX.X | XXX | XXX |
| | XX | | x | | XXX.X | XX.XX | XXX.X | XXX | XXX |

204824

Example : EFF\_T3
Protocol : 204824
Page 1 of n

Population : All Subjects.

Table X
Proportion of Subjects with DGF

Number of Subjects (%)

(N)

Subjects with DGF XXX (%)

204824

: EFF\_T4 : 204824 Page 1 of n Example

Protocol Population : All Subjects.

Table X Proportion of Subjects with Renal Functional Graft within 7 Days after Transplant

Number of Subjects (%)

(N)

| Primary Non DGF | XXX (%) |
|-----------------------------------|---------|
| 3 day Functional DGF | XXX (%) |
| 7 day Functional DGF | XXX (%) |
| 3 day Intermediate Graft Function | XXX (%) |
| 7 day Intermediate Graft Function | XXX (%) |
| 3 day Immediate Graft Function | XXX (%) |
| 7 day Immediate Graft Function | XXX (%) |


Example : EFF\_T5 Protocol : 204824

Population : All Subjects

Table X
Summary of Maximum Emergent QTc Values by Category

Baseline (N = xx)Enhanced Monitoring (N = xx)Mean max Criteria N Mean QTc SD Criteria N SD QTc QT <= 480 msec QTc > 530 msecXXXX.X XX.XX XXXX.X XX.XXQT (uncorr) > 600 msecXXXX.X XX.XXBundle Branch Block with QTc >= 550 msecXXXX.XXX.XX XXXX.XXX.XXQT < =500 msecQT (uncorr) > 600 msec XXXX.X XX.XX

Note: QTc value could be QTcB or QTcF depends on collected data.

204824

Example : SAFE\_L1

Protocol : 204824
Population : All Subjects


Listing X Listing of XXX

| Treatment | Subj. | Analyte (units) | Visit | Actual Date | Planned<br>Relative<br>Time | Time<br>Sample<br>Taken | Result | Change<br>from<br>Baseline |
|---|---|---|---|---|---|---|---|---|
| GSK1070806<br>3mg/kg | PPD | XXX | DAY 1 | PPD | PRE DOSE | 9:48 | 0.9 | |
| - 6 6 | | | DAY 1 | | 4 Hr | 9:48 | 1.10 | 0.20 |
| | | | DAY 29 | | 4 Hr | 9:48 | 2.60 | 1.70 |
| | | | DAY 85 | | 4 Hr | 9:48 | 1.10 | 0.20 |

NOTE: Table adjusted accordingly to the study data.

204824


Example : SAFE\_L2 Protocol : 204824

Protocol : 204824
Population : All Subjects

Listing X

| | _ | | |
|---------------------|--------------------|-----------------------|------|
| Listing of Patients | Hospitalization an | nd Re-hospitalization | Stay |

| Subject | Age/Gender | Race | DGF (Y/N) | Hosp. Date | Discharge Date | Length of Stay (Day) |
|---|---|---|---|---|---|---|
| XXXXXXX | XX/X | XX | X | XX/XX/XXXX | XX/XX/XXXX | XX |
| | | | | XX/XX/XXXX | XX/XX/XXXX | XX |
| XXXXXXX | XX/X | XX | X | XX/XX/XXXX | XX/XX/XXXX | XX |

204824

Example : SAFE\_L3 Protocol : 204824

Population : All Subjects


Table X

Listing of Donor Virology

| Subject | Age/Gender | Race | Virology Type | Positive (yes/no) |
|---------|------------|------|---------------|-------------------|
| XXXXXXX | XX/X | XX | Hepatitis B | |
| | | | Hepatitis C | |
| | | | HIV | |
| | | | EBV | |

204824


Example : SAFE\_L4 Protocol : 204824

Population : All Subjects

Table X Listing of Donor Characteristics

| Subject | Age/Gender | Race | Characteristics | Value |
|---|---|---|---|---|
| XXXXXXX | XX/X | XX | Cold Ischiemic Time | |
| | | | Warm Ischemic Time | |
| | | | Last Creatinine before Transplant | |
| | | | <b>Donor Medical Conditions</b> | |
| | | | Biopsy Performed | Yes/No |
| | | | Transport System | Ice/Perfusion |

204824

Example : SAFE\_L5 Page 1 of X

Protocol : 204824 Population : PK

Table X Listing of Serum IL-18 vs. PK. Plasma Concentrations

| Subject | Age/Gender | Race | Serum IL-18 (drug bound, total or free) | PK Plasma Concentrations |
|---|---|---|---|---|
| XXXXXXX | XX/X | XX | XX.X | XX.X |

#### 11.11. Appendix 11: Summary of Change of Amendment 1

Consistent with the recent protocol amendment, change the number of patients for the dose escalation interim analysis from 8-10 to 6.

The following outputs have been removed from the IA1 delivery as a result of a team decision that these variables are no longer required for a dose escalation decision:

Table 2.11; 2.12; 2.13; 2.14; 2.15; 2.16; 2.17; 2.18; 2.19; 2.20; 2.21; 2.25; 2.26

Figure 2.03; 2.05; 2.06; 2.07; 2.08

Table 4.03

Figure 4.01; 4.02; 4.03; 5.01

ICH listing 3; 9

Non-ICH listing 26; 27; 41